CLINICAL TRIAL: NCT04973358
Title: BUCCOTHERM : Randomized Clinical Trial to Determine the Effect of a Mouthwash on the Preservation of the Ecology of the Oral Microbiome and Its Compatibility With Health
Brief Title: Clinical Trial to Determine the Effect of a Mouthwash on the Preservation of the Ecology of the Oral Microbiome and Its Compatibility With Health
Acronym: BUCCOTHERM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35RC21_9796_BUCCOTHERM; 2021-A01541-40 (Other: N° IDRCB)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: Buccal Microbiota
Keywords: mouthwash

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BuccoTherm (Experimental): buccotherm mouthwash
  Interventions: Other: buccotherm mouthwash
- Placebo (Placebo Comparator): placebo mouthwash
  Interventions: Other: placebo mouthwash

INTERVENTIONS:
Other: buccotherm mouthwash — twice a day for 14 weeks
  Arms: BuccoTherm
Other: placebo mouthwash — twice a day for 14 weeks
  Arms: Placebo

SUMMARY:
The microbiota of the human body is essential to life, and plays an essential role in the protection and development of various pathological conditions. There is a symbiotic or mutualistic relationship between humans and their microbiota. However, when the microbiota becomes dysbiotic, it is associated with pathological conditions. In the oral cavity, dysbiosis is responsible for caries and periodontal pathologies, but other associations have been demonstrated or are suspected with distant pathologies (rheumatoid arthritis, Alzheimer's disease). Mouthwashes are used therapeutically or daily to maintain oral health. The main studies reporting their effects on the ecology of the oral microbiota are for the most part limited to Pasteurian culture techniques (40% of bacteria are not yet cultivable). The advent of new generations of sequencing allows to overcome this limitation and to explore the complexity of bacterial communities, i.e. the symbiosis or dysbiosis of the entire bacterial ecosystem. The control of the oral microbiota to prevent pathologies requires a better knowledge of the oral microbial ecology and will allow the development of new approaches that consider the process of biofilm formation and the disruption of bacterial communication networks. The effects of daily mouthwash must therefore be studied at the level of the entire bacterial community.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older:
* with at least 20 permanent natural teeth, excluding crowns;
* affiliated to a social security system;
* having received information about the protocol and having given their free, informed and written consent.

Exclusion Criteria:

* with periodontitis in the month prior to inclusion;
* with significant carious lesions deeply modifying the oral microbiota in the month prior to inclusion;
* having undergone oral surgical treatment within 3 months prior to inclusion;
* wearing orthodontic appliances;
* having undergone periodontal procedures in the month prior to inclusion;
* suffering from severe chronic pathologies deemed incompatible with study entry;
* allergic to one of the swab components;
* allergic to any of the components of the BUCCOTHERM mouthwash or the placebo;
* on drugs that may cause gingival hypertrophy, such as Hydantoins (phenytoin), Dihydropyridines, Diltiazem or Ciclosporin;
* Medications that can cause gingival bleeding (anticoagulants, antiplatelet agents and aspirin);
* Antibiotic therapy or professional scaling in the month prior to inclusion;
* having used oral or topical antibiotics, antiseptics and/or antifungals (e.g., mouthwash, dental gels, etc.) in the month prior to inclusion.
* Subjects with poor written and spoken French language skills;
* previously included in the BUCCOTHERM study;
* simultaneously participating in another trial that may interfere with the conduct of the BUCCOTHERM study or in a period of exclusion after participation in another clinical study;
* protected persons (adults under legal protection (legal guardianship, curatorship, tutorship), persons deprived of liberty, pregnant or breastfeeding women, women of childbearing age without effective contraception (estrogen-progestin treatments, IUD, tubal ligation), minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Commensal species of the oral microbiota | week 14
  Change from baseline in commensal species at 14 weeks
Alpha and beta diversity of the oral microbiota | week 14
  Change from baseline in alpha and beta diversity at 14 weeks
Coefficient of dysbiosis/symbiosis of the oral microbiota | week 14
  Change from baseline in coefficient of dysbiosis/symbiosis at 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Meuric Vincent, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No